CLINICAL TRIAL: NCT02818517
Title: Evaluation and Management of Cardio Toxicity in Oncologic Patients
Status: Recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, Udi Chorin MD, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-16-UC-0228-16-TLV-CTIL
Record Dates: First submitted 2016-06-15; First posted 2016-06-29 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Angiotensin-Converting Enzyme Inhibitors; Adrenergic beta-Antagonists

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart failure: Evaluating the cardio toxicity effect of chemotherapy and radiation and estimating the effect of ACE inhibitors and beta blockers in the prevention of heart failure.
  Interventions: Other: ACE inhibitors; Other: beta blockers

INTERVENTIONS:
Other: ACE inhibitors — Evaluating the cardio toxicity effect of chemotherapy and radiation and estimating the effect of ACE inhibitors and beta blockers in the prevention of heart failure.
Other: beta blockers — Evaluating the cardio toxicity effect of chemotherapy and radiation and estimating the effect of ACE inhibitors and beta blockers in the prevention of heart failure.

SUMMARY:
The survival rate of cancer patients has greatly increased over the past decades' mainly due to early detection and the use of new medications with higher doses and combined protocols. This achievement comes with the price of cardio toxicity, leading to cardiac dysfunction ranged from transient asymptomatic left ventricular dysfunction to cardiac death. In the long term, the risk of death from cardiovascular causes exceeds that of tumor recurrence for many types of cancer. As a result of the increasing number of long-term cancer survivors the magnitude of this problem is growing. Early identification of cardio toxicity can be identified by clinical follow-up and the use of electrocardiography, cardiac biomarkers (Troponin, brain natriuretic peptide) and echocardiogram. Past studies imply that the addition of angiotensin-converting-enzyme inhibitor (ACE inhibitor) and beta blockers to the patient's treatment may prevent the development of cardiac dysfunction. However, currently there are no specific or clear guidelines for the follow-up and management of cardio-toxicity in cancer patients.

The aim of the study: To try to identify who are the patients at increased risk for developing cardio toxicity, by follow up of clinical evaluation, cardiac biomarkers and echocardiogram examination, in purpose of early diagnosis, management and prevention of cardiac events. For achieving this the investigators will build a registry which will include all the oncologic patients going an evaluation in the cardio-oncology clinic in the Tel Aviv Medical Center .

DETAILED DESCRIPTION:
The survival rate of cancer patients has greatly increased over the past decades' mainly due to early detection and the use of new medications with higher doses and combined protocols. This achievement comes with the price of cardio toxicity, leading to cardiac dysfunction ranged from transient asymptomatic left ventricular dysfunction to cardiac death. In the long term, the risk of death from cardiovascular causes exceeds that of tumor recurrence for many types of cancer. As a result of the increasing number of long-term cancer survivors the magnitude of this problem is growing. Early identification of cardio toxicity can be identified by clinical follow-up and the use of electrocardiography, cardiac biomarkers (Troponin, brain natriuretic peptide) and echocardiogram. Past studies imply that the addition of angiotensin-converting-enzyme inhibitor (ACE inhibitor) and beta blockers to the patient's treatment may prevent the development of cardiac dysfunction. However, currently there are no specific or clear guidelines for the follow-up and management of cardio-toxicity in cancer patients.

The aim of the study: To try to identify who are the patients at increased risk for developing cardio toxicity, by follow up of clinical evaluation, cardiac biomarkers and echocardiogram examination, in purpose of early diagnosis, management and prevention of cardiac events. For achieving this the investigators will build a registry which will include all the oncologic patients going an evaluation in the cardio-oncology clinic in the Tel Aviv Medical Center .

The study will be composed of two groups:

1. The retrospective group analysis will include all oncologic patients who were evaluated in the cardio-oncology clinic between 01 January 2014 until 31 May 2016.
2. The prospective group will include all oncologic patients who will be evaluated in the cardio-oncology clinic from 01 June 2016 onward.

The patients will sign an informed consent form. The data collected will include demographic: gender, age, duration of hospitalization, diagnosis, symptoms, clinical as well as laboratory, echocardiographic and echicardiogram findings.

The study will be based on unidentified data taken from medical records or medical files of patients. Identified details will be separated in a way that won't enable to review them . All data handling and the separation of the identified data will be done by the Principal Investigator, or sub-investigator in this study, who is in charge of the hearing screening program in Tel Aviv Medical Center.

The study population will include all patients evaluated in the cardio-oncology clinic in our hospital with the diagnosis of cancer and are planned for chemotherapy and/or radiation treatment.

The data collected will include gender, age, cardiovascular risk factors, cardiovascular disease, type of cancer, type of chemotherapy and/or radiation planned, past chemotherapy and/or radiation, vital signs, basic ECG, blood test pre and post therapy (including troponin, CPK, BNP, glucose HBA1C, cholesterol, triglycerides, CRP, WBC, neutrophil count, lymphocyte count, RDW, BNP), Echo at baseline and post therapy (Systolic and diastolic function, strain and valvular function), ACE inhibitor and beta blocker treatment, complication and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patient evaluated in the cardio-oncology clinic in Tel Aviv MC

Exclusion Criteria:

* In the prospective Study - patients not sign an informed consent form.

Exclusion criteria experiment:

Patient reluctance to continue the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be composed of two groups:
  1. The retrospective group analysis will include all oncologic patients who were evaluated in the cardio-oncology clinic between 01 January 2014 until 31 May 2016.
  2. The prospective group will include all oncologic patients who will be evaluated in the cardio-oncology clinic from 01 June 2016 onward.
  The patients will sign an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
ECho-global strain | 2 years
  Predictor of reduction Ejection Fraction
Troponin (ng/ml) | 2 years
  Predictor of reduction Heart failure
ACE inhibitor and beta blocker treatment | 2 years
  estimating the effect of ACE inhibitors and beta blockers preventive treatment for heart failure due to chemotherapy.
BNP (PG/ML) | 2 years
  Predictor of reduction Heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Udi Chorin, MD, Principal Investigator — Tel Aviv MC
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shamai S, Rozenbaum Z, Merimsky O, Derakhshesh M, Moshkovits Y, Arnold J, Topilsky Y, Arbel Y, Laufer-Perl M. Cardio-toxicity among patients with sarcoma: a cardio-oncology registry. BMC Cancer. 2020 Jun 30;20(1):609. doi: 10.1186/s12885-020-07104-9. PMID 32605637